CLINICAL TRIAL: NCT07343414
Title: Impact of Anesthesia Method on Surgical View and Surgeon Satisfaction During Shoulder Arthroscopy: A Prospective Observational Study
Brief Title: Effect of Anesthesia Technique on Surgical View in Shoulder Arthroscopy
Status: Not yet recruiting | Type: Observational
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Harun Tolga Duran, Medical Doctor, Amasya University
Other Study IDs: 2025000139-3
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Arthroscopy; Interscalene Nerve Block; Surgical View Quality; Surgeon Satisfaction
Keywords: Shoulder Arthroscopy; Surgeon Satisfaction; Surgical View Quality; Interscalene Nerve Block; Rotator Cuff Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Anesthesia Group: Patients undergoing elective shoulder arthroscopy who receive general anesthesia as determined by routine clinical practice and patient preference.
- Regional Anesthesia Group: Patients undergoing elective shoulder arthroscopy who receive regional anesthesia [interscalene nerve block/superficial cervical block] combined with sedation as determined by routine clinical practice and patient preference.

SUMMARY:
This prospective observational study evaluates the effect of the anesthesia method (general anesthesia versus regional anesthesia [interscalene nerve block/superficial cervical block] with sedation) on the operating clarity of the surgical view and the surgeon's satisfaction during elective shoulder arthroscopy. The study investigates how these different anesthesia techniques influence intraoperative conditions, specifically bleeding amounts and the visibility of the surgical field, which are critical for the success of this minimally invasive procedure. Additionally, the research will monitor patient-centered outcomes, including postoperative pain levels, recovery time, and potential side effects such as nausea or vomiting, to determine which anesthesia strategy provides the optimal balance of surgical efficiency and patient comfort.

DETAILED DESCRIPTION:
Shoulder arthroscopy is a minimally invasive surgical procedure where the clarity of the surgeon's visual field is critical for technical success and operative efficiency. The quality of the intraoperative view is heavily influenced by perioperative variables, particularly intraoperative bleeding and hemodynamic stability. Consequently, the anesthetic management strategy-whether General Anesthesia (GA) or Regional Anesthesia (RA) [interscalene nerve block/superficial cervical block] combined with sedation-may significantly alter these conditions. This study aims to prospectively evaluate and compare how these two distinct anesthesia methods impact the clarity of the surgical field, and the operating surgeon's satisfaction.

This is a prospective, observational cohort study will conducted at the Sabuncuoğlu Serefeddin Training and Research Hospital. The study utilizes a naturalistic, non-randomized design. There is no interference with the choice of anesthesia; group assignment is determined solely by routine clinical decision-making and patient preference during the preoperative assessment. Patients are recruited and observationally assigned to one of two cohorts based on the technique administered:

* General Anesthesia Group: Patients who elect or are clinically selected to receive general anesthesia.
* Regional Anesthesia Group: Patients who elect or are clinically selected to receive an interscalene nerve block/superficial cervical block combined with sedation.

Intraoperative physiological variables, including heart rate, systolic and diastolic blood pressure, oxygen saturation, and respiratory rate, will be continuously monitored throughout the procedure. The study will also record the feasibility of implementing controlled hypotension and analyze its correlation with intraoperative bleeding amounts. To provide a holistic comparison between anesthesia methods, the study will track postoperative recovery metrics, including the total duration of surgery and anesthesia. Additionally, postoperative pain will be assessed using the Numeric Rating Scale (NRS) at 1, 2, 4, 8, 16, and 24 hours post-procedure. The incidence of opioid-related side effects, such as nausea and vomiting, will be monitored and recorded during the postoperative period .

Primary Assessment:

- Surgical View Evaluation: The clarity of the surgical field and the extent to which bleeding obscures visualization are evaluated using a 5-point Likert scale (1 = Poor/No Visualization: Severe bleeding that completely obscures the field; surgery is extremely difficult or impossible without constant suction/lavage; 2 = Fair Visualization: Significant bleeding obscuring the field; frequent suction/lavage is required to proceed; 3 = Moderate Visualization: Moderate bleeding; the anatomy is visible, but occasional suction/lavage is needed to maintain a clear view; 4 = Good Visualization: Mild bleeding; the surgical field is clear with only rare need for suction/lavage; 5 = Excellent/Crystal Clear Visualization: No significant bleeding; the surgical field is perfectly clear throughout the procedure.)

Sample Size: Based on a preliminary analysis conducted at our center, a distinct difference in the primary outcome (Surgical view evaluation) was observed between the two groups (RA: 3.1 ± 1.2 vs. GA: 4.0 ± 1.5). To detect this difference with a Power (1-beta) of 0.80 and an alpha error of 0.05, a sample size of 37 patients per group is required. Accounting for a 10% dropout rate, the study will enroll a total of 82 patients (41 in the GA group and 41 in the RA group).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 18 to 75 years.
* Patients scheduled for elective shoulder arthroscopy.
* Patients with an ASA (American Society of Anesthesiologists) physical status score of I, II, or III.
* Patients capable of providing informed consent.

Exclusion Criteria:

* Previous surgical procedure performed on the same shoulder.
* Presence of medical contraindications that could affect the choice of anesthesia (coagulopathy, active infection, severe pulmonary diseases)
* Known allergy to local anesthetics or general anesthesia agents
* History of opioid dependence or chronic pain syndrome
* Presence of neurological disorders, particularly those involving the brachial plexus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18 to 75 years) who are scheduled to undergo elective shoulder arthroscopy at the Sabuncuoğlu Şerefeddin Training and Research Hospital. These participants are recruited from the patient pool presenting to the Orthopedics and Traumatology clinic for surgical treatment of shoulder pathologies (rotator cuff tears or impingement). Participants include individuals with an ASA physical status of I, II, or III who are capable of providing informed consent .
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Surgical View Clarity Score | Intraoperative (assessed immediately upon completion of wound closure)
  The clarity of the surgical field and the extent to which bleeding obscures visualization are evaluated by the surgeon using a 5-point Likert scale. The scale ranges from 1 (Poor/No Visualization) to 5 (Excellent/Crystal Clear Visualization).

SECONDARY OUTCOMES:
Surgeon Satisfaction Score | Intraoperative (assessed immediately upon completion of wound closure)
  The operating surgeon's overall satisfaction with the procedure and the conditions provided by the anesthesia is assessed using a 5-point Likert scale. The scale is defined as: 1 = Very Dissatisfied, 2 = Dissatisfied, 3 = Neutral, 4 = Satisfied, 5 = Very Satisfied.
Intraarticular Bleeding Severity | Intraoperative
  The operating surgeon's subjective assessment of the amount of bleeding within the joint during the arthroscopy. This is evaluated using a categorical scale:
  * Good: Minimal bleeding that does not interfere with the procedure.
  * Moderate: Bleeding is present but manageable; does not significantly hinder the procedure.
  * Poor: Significant bleeding that obscures the surgical field and complicates the procedure.
Feasibility of Controlled Hypotension | Intraoperative
  Binary assessment of whether controlled hypotension (systolic blood pressure reduction to reduce bleeding) was successfully applied and maintained during the surgery (Yes/No).
Duration of Surgery | Intraoperative
  The time in minutes measured from the start of the incision to the completion of wound closure.
Duration of Anesthesia | Intraoperative
  The total time in minutes from the induction of anesthesia to the cessation of anesthetic effects/emergence.
Postoperative Pain Score (NRS) | Postoperative hours 1, 2, 4, 8, 16, and 24
  Assessment of patient pain intensity using the Numeric Rating Scale (NRS), where 0 represents "no pain" and 10 represents "worst pain imaginable."
Incidence of Opioid-Related Side Effects | Postoperative 24 hours
  The occurrence of specific side effects associated with opioid use, including nausea, vomiting, and pruritus (itching).
Patient Satisfaction Score | Postoperative 24 hours
  The patient's self-reported level of satisfaction with the perioperative process and their comfort level. This is assessed using a 5-point Likert scale (1 = Very Dissatisfied; 2 = Dissatisfied; 3 = Neutral; 4 = Satisfied; 5 = Very Satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Salih Tüzen, M.D., Principal Investigator — Izmir Katip Celebi University Atatürk Training and Research Hospital
Locations (1):
- Amasya University Sabuncuoglu Serefeddin Educational and Research Hospital, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No